CLINICAL TRIAL: NCT00343733
Title: A 12-Week Open-Label Study With 3 Within-Patient Double-Blind Placebo-Controlled Periods to Evaluate the Efficacy and Safety of OraVescent Fentanyl Citrate Treatment for the Management of Breakthrough Pain in Opioid-Tolerant Patients With Noncancer-Related Chronic Pain
Brief Title: Study to Evaluate the Efficacy and Safety of OraVescent Fentanyl Citrate Treatment for the Management of Breakthrough Pain in Opioid-Tolerant Patients With Noncancer-Related Chronic Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: C25608/3052/BP/US
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Pain
Keywords: diabetic peripheral neuropathy; postherpetic neuralgia; traumatic injury; complex regional pain syndrome; back pain; neck pain; fibromyalgia; chronic pancreatitis; osteoarthritis
MeSH Terms: conditions — Pain; Neuralgia, Postherpetic; Wounds and Injuries; Complex Regional Pain Syndromes; Back Pain; Neck Pain; Fibromyalgia; Pancreatitis, Chronic; Osteoarthritis

INTERVENTIONS:
Drug: OraVescent Fentanyl

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of OraVescent fentanyl treatment compared to placebo treatment monthly over a 12-week treatment period in alleviating breakthrough pain (BTP) in opioid-tolerant patients with noncancer-related chronic pain.

ELIGIBILITY:
Inclusion Criteria:

Patients are included in the study if all of the following criteria are met:

* The patient is willing to provide written informed consent to participate in this study.
* The patient is 18 through 80 years of age.
* Women must be surgically sterile, 2 years postmenopausal, or, if of childbearing potential, using a medically accepted method of birth control (ie, barrier method with spermicide, steroidal contraceptive [oral, transdermal, implanted, and injected contraceptives must be used in conjunction with a barrier method], or intrauterine device [IUD]) and agree to continued use of this method for the duration of the study.
* The patient has chronic pain of at least 3 months' duration associated with any of the following conditions: diabetic peripheral neuropathy, postherpetic neuralgia, traumatic injury, complex regional pain syndrome, back pain, neck pain, fibromyalgia (documented diagnosis), chronic pancreatitis, or osteoarthritis. Other chronic painful conditions may be evaluated for entry upon discussion with, and written approval from, the Cephalon Medical Monitor.
* The patient is currently using 1 of the following: at least 60 mg of oral morphine/day, or at least 25 mcg of transdermal fentanyl/hour, or at least 30 mg of oxycodone/day, or at least 8 mg of hydromorphone/day, or an equianalgesic dose of another opioid/day as a stable dose of ATC therapy for at least the previous 30 days prior to enrollment in the study.
* The patient reports an average pain intensity score, over the prior 24 hours, of 6 or less (0=no pain through 10=worst pain) for his/her chronic pain.
* The patient experiences, on average, 1 to 4 BTP episodes (defined as temporary flares of severe or excruciating pain) per day while taking ATC opioid therapy, and on average, the duration of each BTP episode is less than 4 hours.
* The patient currently uses opioid therapy for alleviation of BTP episodes, occurring at the location of the chronic pain, and achieves at least partial relief.
* The patient is able to effectively self-administer the study drug and complete the electronic diary.

Exclusion Criteria:

Patients are excluded from participating in this study if 1 or more of the following criteria are met:

* The patient has uncontrolled or rapidly escalating pain as determined by the investigator (ie, the ATC therapy may be expected to change between the first and last treatments with study drug), or has pain uncontrolled by therapy that could adversely impact the safety of the patient or that could be compromised by treatment with study drug.
* The patient has known or suspected hypersensitivities, allergies, or other contraindications to any ingredient in the study drug.
* The patient has a recent history (within 5 years) or current evidence of alcohol or other substance abuse.
* The patient has cardiopulmonary disease that would, in the opinion of the investigator, significantly increase the risk of treatment with potent synthetic opioids.
* The patient has medical or psychiatric disease that, in the opinion of the investigator, would compromise collected data.
* The patient is expected to have surgery during the study and it is anticipated that the surgery will alleviate the patient's pain.
* The patient has had therapy before study drug treatment that, in the opinion of the investigator, could alter pain or response to pain medication.
* The patient is pregnant or lactating.
* The patient has participated in a previous study with OraVescent fentanyl.
* The patient has participated in a study involving an investigational drug in the previous 30 days.
* The patient has received a monoamine oxidase inhibitor (MAOI) within 14 days before the first treatment with study drug.
* The patient has any other medical condition or is receiving concomitant medication/therapy (eg, regional nerve block) that would, in the opinion of the investigator, compromise the patient's safety or compliance with the study protocol, or compromise collected data.
* The patient is involved in active litigation in regard to the chronic pain currently being treated.
* The patient has a positive urine drug screen (UDS) for a medication not prescribed by the physician currently treating the chronic pain.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2006-08; Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
The primary objective is to evaluate the efficacy of OraVescent fentanyl treatment compared with placebo treatment following 12 weeks of treatment in alleviating breakthrough pain (BTP) in opioid-tolerant patients with noncancer-related chronic pain.

CONTACTS AND LOCATIONS:
Locations (21):
- United States (21):
  - Hot Springs Pain Clinic, Hot Springs, Arkansas
  - Samaritan Center for Medical, Los Gatos, California
  - Pacific Neuroscience Medical Group, Inc., Oxnard, California
  - Centre for Rheumatology, Fort Lauderdale, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Atlas Research, Orlando, Florida
  - Gold Coast Research, LLC, Plantation, Florida
  - Comprehensive Pain Care, PC, Marietta, Georgia
  - Drug Studies America, Marietta, Georgia
  - Best Clinical Trials, Inc., New Orleans, Louisiana
  - Best Clinical Trials, LLC, New Orleans, Louisiana
  - Brigham Women's Hospital, Boston, Massachusetts
  - Pain Management Associates, Independence, Missouri
  - Montana Neuroscience Institute, Missoula, Montana
  - Lovelace Scientific Resources, Albuquerque, New Mexico
  - Five Towns Neuroscience Research, Lawrence, New York
  - PharmQuest, Greensboro, North Carolina
  - Center for Clinical Research, Winston-Salem, North Carolina
  - Legacy Emanuel Pain Management, PC, Portland, Oregon
  - Clinical Research Center, West Reading, Pennsylvania
  - Advanced Pain Management, Virginia Beach, Virginia